CLINICAL TRIAL: NCT06103110
Title: Effect of Order and Conjugation of Different Photobiomodulation Therapies and Anterior Repositioning Appliance in Management of TMD Cases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Mohamed shady, Assistant Professor, Mansoura University
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: A04100522
Record Dates: First submitted 2023-10-22; First posted 2023-10-26 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: TMJ Disorder
MeSH Terms: conditions — Temporomandibular Joint Disorders | interventions — Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- anterior repositioning appliance followed by Infra-red LED therapy (Experimental): anterior repositioning appliance followed by Infra-red LED therapy
  Interventions: Device: Photobiomodulation
- Infra-red LED therapy followed by anterior repositioning appliance (Experimental): Infra-red LED therapy followed by anterior repositioning appliance
  Interventions: Device: Photobiomodulation
- anterior repositioning appliance followed by Low level Laser therapy (Experimental): anterior repositioning appliance followed by Low level Laser therapy
  Interventions: Device: Photobiomodulation
- Low level Laser therapy followed by anterior repositioning appliance (Experimental): Low level Laser therapy followed by anterior repositioning appliance
  Interventions: Device: Photobiomodulation

INTERVENTIONS:
Device: Photobiomodulation — Laser therapy using low level laser

SUMMARY:
This study aimed to evaluate the effect of using Low level laser therapy / Infrared led therapy with anterior repositioning appliance in anterior dislocation patients with reduction (ADDwR) concerning:

1. Range of mandibular motion
2. Helkimo questioner to evaluate :

A -TMJ function B -Muscle pain C -TMJ pain D - Pain on movement of the mandible

Four groups created randomly each 10 patients as following:-

Group 1: anterior repositioning appliance followed by Infra-red LED therapy Group 2: Infra-red LED therapy followed by anterior repositioning appliance Group 3: anterior repositioning appliance followed by Low level Laser therapy Group4: Low level Laser therapy followed by anterior repositioning appliance

Evaluation was done through the following methods

Clinical examination:

1. A detailed questionnaire by the examiner was recorded for each patient including: personal data, chief complaint, medical as well as past dental histories
2. Magnetic resonance imaging (MRI) for each patient, the clinical diagnosis of disc displacement with reduction confirmed by MRI.
3. Maximum inter-incisal opening (MIO):was measured by Vernier caliper in millimetres (mm) as the vertical distance between the incisal edges of maxillary and mandibular central incisors.
4. Range of lateral mandibular excursions was also measured using Vernier caliper in millimetres as the horizontal distance extending from maxillary midline to mandibular midline. This was measured by asking the patient to move the mandible to one side then to the other side to the maximum extent.
5. Helkimos clinical dysfunction scale.

DETAILED DESCRIPTION:
This study included forty patients suffering from TMJ internal derangement with reduction. They were all selected from the outpatient clinic of the Prosthodontics Department, Faculty of Dentistry, Mansoura University. All the included patients showed persistent restriction of mouth opening as well as TMJ pain and clicking. Patients suffering from inflammatory or connective tissue diseases, neurologic disorders, history of bony or ibrous adhesion, gross mechanical restrictions and condylar fractures, previous TMJ surgery, TMJ ankylosis, or acute infection were all excluded. Moreover, muscle relaxants, non-steroidal anti-inflammatory drugs within 48 h preoperatively, corticosteroid injection at treatment site within one month or systemic use of corticosteroids within 2 weeks were also excluded in this study.

Clinical examination:

1. A detailed questionnaire by the examiner was recorded for each patient including: personal data, chief complaint, medical as well as past dental histories
2. Magnetic resonance imaging (MRI) for each patient, the clinical diagnosis of disc displacement with reduction was confirmed by MRI.
3. Maximum inter-incisal opening (MIO):was measured by Vernier caliper in millimetres (mm) as the vertical distance between the incisal edges of maxillary and mandibular central incisors.
4. Range of lateral mandibular excursions was also measured using Vernier caliper in millimetres as the horizontal distance extending from maxillary midline to mandibular midline. This was measured by asking the patient to move the mandible to one side then to the other side to the maximum extent.
5. Helkimos clinical dysfunction scale.

Four groups created randomly each 10 patients as following:-

Group 1: anterior repositioning appliance followed by Infra-red LED therapy Group 2: Infra-red LED therapy followed by anterior repositioning appliance Group 3: anterior repositioning appliance followed by Low level Laser therapy Group4: Low level Laser therapy followed by anterior repositioning appliance

Anterior Repositioning Appliance

This appliance, is to alter the maxillomandibular relationship so that a more anterior position assumed by the mandible. Acrylic guiding ramp added to the anterior third of the maxillary appliance that direct the mandible into a more forward position, upon closing. This type of appliance designed to be used in treating patients with anterior disk displacement with reduction. It was supposed that by altering the mandibular position in this manner, the anteriorly displaced disks could return back to its normal position (recaptured).

LOW LEVEL LASER APPLICATION The LLLT were applied bilaterally to the face, five points were irradiated: three points around the TMJ, one point on the temporalis and one on the masseter. The treatment was performed twice a week for three consecutive weeks

INFRA RED LED APPLICATION The LED therapies were applied bilaterally to the face for 60 s/point. Five points were irradiated: three points around the TMJ, one point on the temporalis and one on the masseter. Eight sessions of the phototherapy were performed, twice a week for 4 weeks

Follow up:

Patients were re-examined for maximum openening ,lateral movement and Helkimos scale after 6 months.

ELIGIBILITY:
Inclusion Criteria:

* suffering from TMJ internal derangement with reduction.
* All the included patients show persistent restriction of mouth opening as well as TMJ pain and clicking.

Exclusion Criteria:

* Patients suffering from inflammatory or connective tissue diseases,
* neurologic disorders
* history of bony or fibrous adhesion
* gross mechanical restrictions and condylar fractures
* previous TMJ surgery
* TMJ ankylosis
* acute infection
* muscle relaxants, non-steroidal anti-inflammatory drugs within 48 h preoperatively, corticosteroid injection at treatment site within one month or systemic use of corticosteroids within 2 weeks

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2022-10-20 (Actual); Primary Completion 2023-06-24 (Actual); Study Completion 2023-08-03 (Actual)

PRIMARY OUTCOMES:
Range of motion | Before treatment (T0) , After 6 months (T6)
  Maximum opening, lateral movement and protrusion

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura University, Faculty of dentistry, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: No